CLINICAL TRIAL: NCT02176473
Title: Evaluating the Feasibility and Efficacy of Computerized Cognitive Behavioral Therapy in Prolonging the Antidepressant Effects of Electroconvulsive Therapy
Brief Title: Computerized Cognitive Behavioral Therapy and Electroconvulsive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1404013837
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Computerized Cognitive Behavioral Therapy (Experimental): A computerized version of CBT has been developed in an effort to more widely disseminate the powerful effects of this psychotherapy modality, with studies showing efficacy comparable to that of traditional CBT.8 The present study aims to further investigate the feasibility of combining ECT and computerized CBT (c-CBT).
  Interventions: Behavioral: Computerized Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Computerized Cognitive Behavioral Therapy — The c-CBT software focuses on the same principles of traditional CBT, namely, "identifying, labeling, and modifying automatic thoughts; the link between thought and action; identifying and modifying schemas; and identifying and correcting cognitive errors."9 C-CBT is delivered in 9 online lessons, each designed to take 30-45 minutes to complete. The software provides modeling of CBT principles (in the form of short videos), enables an interactive forum by giving users feedback based on responses to questions, and encourages participants to employ the skills learned in CBT to their situations. A 9-minute video demonstrating the functionality of Good Days Ahead can be found at: http://www.empower-interactive.com/solutions/good-days-ahead/.

SUMMARY:
In an open-label feasibility study, fifteen will be recruited to participate in the study from among those who have already chosen of their own accord to undergo ECT (standard of care) at Yale Psychiatric Hospital for treatment of a depressive episode. These patients will receive computer-assisted cognitive behavior therapy (CCBT).

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* meet DSM-5 criteria for depressive episodes
* able to use a computer

Exclusion Criteria:

* diagnosis of an axis II (personality disorder)
* active suicidal thoughts with a plan
* current substance use disorder
* non-affective psychosis
* prior treatment with ECT in the past 6 months
* CBT treatment in the past 12 months
* dementia
* delirium or another other neurological or mental disease that might affect cognition or the ability to meaningfully participate in computerized CBT

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | Baseline
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression .
  The treatment group will undergo depression rating scales (as well as cognitive screening) at baseline, at 2 weeks during their index course of ECT, following the completion of the ECT phase, and then every 5 weeks for a total of 25 weeks total after the completion of the ECT phase. Depression rating scales will include the BDI, QIDS-SR, MADRS, CGI, and MOCA. During the 10 weeks of their c-CBT course, they will also complete self-rating scales on a more frequent basis (every 2.5 weeks); these scales are the BDI and QIDS-SR.
Beck Depression Inventory | week 2
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression .
  The treatment group will undergo depression rating scales (as well as cognitive screening) at baseline, at 2 weeks during their index course of ECT, following the completion of the ECT phase, and then every 5 weeks for a total of 25 weeks total after the completion of the ECT phase. Depression rating scales will include the BDI, QIDS-SR, MADRS, CGI, and MOCA. During the 10 weeks of their c-CBT course, they will also complete self-rating scales on a more frequent basis (every 2.5 weeks); these scales are the BDI and QIDS-SR.
Beck Depression Inventory | Week 5 through week 15
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression .
  The treatment group will undergo depression rating scales (as well as cognitive screening) at baseline, at 2 weeks during their index course of ECT, following the completion of the ECT phase, and then every 5 weeks for a total of 25 weeks total after the completion of the ECT phase. Depression rating scales will include the BDI, QIDS-SR, MADRS, CGI, and MOCA. During the 10 weeks of their c-CBT course, they will also complete self-rating scales on a more frequent basis (every 2.5 weeks); these scales are the BDI and QIDS-SR.

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomology (QIDS) | Baseline, Week 2, week 5, week 10, week 15
  The16 item Quick Inventory of Depressive Symptomatology (QIDS) (an abbreviated version of the 30 item Inventory of Depressive Symptomatology (IDS) is designed to assess the severity of depressive symptoms.
  The treatment group will undergo the same depression rating scales (as well as cognitive screening) at baseline, at 2 weeks during their index course of ECT, following the completion of the ECT phase, and then every 5 weeks for a total of 25 weeks total after the completion of the ECT phase. During the 10 weeks of their c-CBT course, they will also complete self-rating scales on a more frequent basis (every 2.5 weeks); these scales are the BDI and QIDS-SR.
Montgomery-Åsberg Depression Rating Scale ( MADRS) | Baseline, Week 2, week 5, week 10, week 15
  The Montgomery-Åsberg Depression Rating Scale ( MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders.
  The treatment group will undergo the same depression rating scales (as well as cognitive screening) at baseline, at 2 weeks during their index course of ECT, following the completion of the ECT phase, and then every 5 weeks for a total of 25 weeks total after the completion of the ECT phase. During the 10 weeks of their c-CBT course, they will also complete self-rating scales on a more frequent basis (every 2.5 weeks); these scales are the BDI and QIDS-SR.
Clinical Global Impression (CGI) | Baseline, Week 2, week 5, week 10, week 15
  The Clinical Global Impression rating scales are commonly used measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders.
  The treatment group will undergo the same depression rating scales (as well as cognitive screening) at baseline, at 2 weeks during their index course of ECT, following the completion of the ECT phase, and then every 5 weeks for a total of 25 weeks total after the completion of the ECT phase. During the 10 weeks of their c-CBT course, they will also complete self-rating scales on a more frequent basis (every 2.5 weeks); these scales are the BDI and QIDS-SR.
Montreal Cognitive Assessment (MoCA) | Baseline, Week 2, week 5, week 10, week 15
  The Montreal Cognitive Assessment (MoCA) measures mild cognitive impairment.
  The treatment group will undergo the same depression rating scales (as well as cognitive screening) at baseline, at 2 weeks during their index course of ECT, following the completion of the ECT phase, and then every 5 weeks for a total of 25 weeks total after the completion of the ECT phase. During the 10 weeks of their c-CBT course, they will also complete self-rating scales on a more frequent basis (every 2.5 weeks); these scales are the BDI and QIDS-SR.

CONTACTS AND LOCATIONS:
Overall Officials: Samule Wilkonson, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States